CLINICAL TRIAL: NCT04384276
Title: Simplifying Home Weight Monitoring for Infants With Cleft Lip and/or Palate Differences to Determine if Use of an In-home Scale Leads to Better Compliance With Weight Monitoring Recommendations
Brief Title: Weigh Easy: Simplifying Home Weight Monitoring for Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shao Jiang, Plastic Surgeon, Children's Mercy Hospital Kansas City
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: STUDY00000822
Record Dates: First submitted 2020-02-06; First posted 2020-05-12 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Cleft Lip and Palate
Keywords: Weight Monitoring
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Intervention Model Description: A single experimental group will be enrolled prospectively to use the Weigh Easy system. Due to the potential impacts of weight gain within this patient population and the lifelong implications of early malnutrition, we do not feel we can safely randomize a prospective control group. As a result, a retrospective control group will be enrolled to enable a comparison of outcomes between those families using the Weigh Easy system and those who did not. All patients, both retrospective and prospective, will be treated according to the standard cleft lip and/or palate treatment protocols and followed by the registered nutritionists who routinely participate in the Cleft and Craniofacial Clinic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective Weigh Easy (Experimental): Patients enrolled onto this arm of the study will use the Weigh Easy system for weight tracking in the first three months of life. Weights will be measured in home using the Weigh Easy scale and transmitted to the study team via the Weigh Easy eClipboard message. A notification scheme will be activated for weights found to have plateaued or decreased to ensure that the infant's standard of care nutritionist and provider are able to follow up and recommend additional interventions to counteract the weight change.
  After three months, families will complete a satisfaction survey to determine if the Weigh Easy system was preferable or if there are any improvements that could be made.
  All other aspects of the patients' care will follow the standard of care for cleft and craniofacial diagnoses and will be guided by the nutritionists specializing in cleft and craniofacial care.
  Interventions: Other: The Weigh Easy System
- Retrospective Control Arm (Other): Patients enrolled onto the control arm will have retrospectively presented to the Cleft and Craniofacial Clinic from January 1, 2016 to December 31, 2018 as infants. These patients were treated with the standard of care for cleft and craniofacial diagnoses and were followed by the nutritionists specializing in cleft and craniofacial care.
  Interventions: Other: Retrospective Control

INTERVENTIONS:
Other: The Weigh Easy System — By use of a small user-friendly luggage scale, the family can easily and safely obtain a weight within the comfort of their own home. Using the Weigh Easy eClipboard, a message will be sent to the family on a weekly basis via Cerner's Message Center that will include a link. The link will be used by parents to enter and submit the patient's current weight. Upon submission, the weight will be transmitted into the patient's EMR after it's reviewed and accepted by a member of the study team. When the weight is received in the system, an alert will be triggered that will notify the study team of its arrival. While the Weigh Easy eClipboard function does qualify as a device, as the investigators will be making clinical decisions based off of the data received through the form, the device is not being used investigationally on this study. The eClipboard function is a standard part of the Cerner framework and has been previously investigated and vetted by for safety and efficacy.
  Arms: Prospective Weigh Easy
Other: Retrospective Control — No interventions will be administered to the historical control group.
  Arms: Retrospective Control Arm

SUMMARY:
This single-site, experimental, pilot study in infants identified from 0 - 3 months of age who present to the Cleft and Craniofacial Clinic with a cleft lip and/or palate will compare weight outcomes of infants who used the Weigh Easy system to monitor weight and historical infants whose weights were monitored without the Weigh Easy system.

DETAILED DESCRIPTION:
Patients will be recruited at the earliest possible visit to the Cleft and Craniofacial Clinic. At this visit, families will complete the consent process. After consent is obtained, the study team will ensure that the family is signed up for the Patient Portal and will provide a demonstration of how to safely obtain a weight using the Weigh Easy scale and the infant's car seat. In addition to the luggage scale, a handout will also be sent home with the family, including instructions and safety tips for weighing their infant and instructions for submitting a weight via the Patient Portal.

Families will be asked to submit a weight, obtained with the Weigh Easy scale, via the Weigh Easy eClipboard message on a weekly basis for 3 months.

Three months after the family is enrolled onto the study, the family will be provided the Parental Satisfaction Survey to complete. This will occur at a clinic visit, in the event that a standard of care visit occurs within the window for the visit. If a clinic visit is unavailable, the surveys will be emailed to the family and three reminders will be sent if the survey is not completed in a timely manner.

ELIGIBILITY:
Prospective Group:

Inclusion Criteria:

* Newborn patient ≤ 12 weeks old
* Referred to Children's Mercy Hospital Multidisciplinary Cleft Team from December 1, 2019 - November 30, 2020
* With a diagnosis of cleft lip and/or cleft palate
* Male or female infant of any ethnic background

Exclusion Criteria:

* Infant with secondary major birth defect such as heart or abdominal wall defect in addition to cleft condition
* Infant who is placed in foster care prior to or during the applicable study period
* Patient parents unable to complete an electronic survey.
* Patient parents unable to speak and read Spanish or English.

Retrospective Group:

Inclusion Criteria:

* Newborn patient ≤ 12 weeks old
* Referred to Children's Mercy Hospital Multidisciplinary Cleft Team from January 1, 2016 to June 30, 2019
* With a diagnosis of cleft lip and/or cleft palate
* Male or female infant of any ethnic background

Exclusion Criteria:

* Infant with secondary major birth defect such as heart or abdominal wall defect in addition to cleft condition

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Weight | up to 3 months
  Weight will be recorded for the duration of the study to identify points of weight destabilization.
Change in Nutritional Interventions | up to 3 months
  Recommended nutritional interventions will be recorded and analyzed against the recorded weights to identify any correlations to improved growth.
Change in Admissions | up to 3 months
  Number of admission due to feeding problems or failure to thrive will be analyzed by comparing the number and frequency of admissions between the retrospective and prospective cohorts.

SECONDARY OUTCOMES:
Parental Satisfaction: survey | Month 3
  The Weigh Easy Parental Satisfaction Survey will be used to create a satisfaction score for each family participating. Answers to this survey will be built using a five-point Likert scale. Minimum score: 4, Maximum score: 20, with higher scores indicating lower parental satisfaction. The survey will be administered at a standard of care appointment three months after enrollment (± 1 month) or via email if an appointment is unavailable during this window. This variable will be measured for the prospective cohort only.

CONTACTS AND LOCATIONS:
Overall Officials: Shao Jiang, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- The Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual patient data only can be shared with other researchers, however the necessary contracting will be needed prior to any data can be shared.

REFERENCES:
- [Background] Avedian LV, Ruberg RL. Impaired weight gain in cleft palate infants. Cleft Palate J. 1980 Jan;17(1):24-6. PMID 6928113
- [Background] Barrett, D. E., Radke-Yarrow, M., & Klein, R. E. (1982). Chronic malnutrition and child behavior: Effects of early caloric supplementation on social and emotional functioning at school age. Developmental Psychology, 18(4):541-556. doi:10.1037/0012-1649.18.4.541
- [Background] Beaumont D. A study into weight gain in infants with cleft lip/palate. Paediatr Nurs. 2008 Jul;20(6):20-3. doi: 10.7748/paed2008.07.20.6.20.c6626. PMID 18686410
- [Background] Gregory KE, Radovinsky L. Research strategies that result in optimal data collection from the patient medical record. Appl Nurs Res. 2012 May;25(2):108-16. doi: 10.1016/j.apnr.2010.02.004. Epub 2010 Apr 9. PMID 20974093
- [Background] Hartley SL, MacLean WE Jr. A review of the reliability and validity of Likert-type scales for people with intellectual disability. J Intellect Disabil Res. 2006 Nov;50(Pt 11):813-27. doi: 10.1111/j.1365-2788.2006.00844.x. PMID 16999781
- [Background] Idohou-Dossou N, Wade S, Guiro AT, Sarr CS, Diaham B, Cisse D, Beau JP, Chappuis P, Hoffman D, Lemonnier D. Nutritional status of preschool Senegalese children: long-term effects of early severe malnutrition. Br J Nutr. 2003 Dec;90(6):1123-32. doi: 10.1079/bjn2003990. PMID 14641972
- [Background] Jones WB. Weight gain and feeding in the neonate with cleft: a three-center study. Cleft Palate J. 1988 Oct;25(4):379-84. PMID 3060285
- [Background] Kaye A, Thaete K, Snell A, Chesser C, Goldak C, Huff H. Initial Nutritional Assessment of Infants With Cleft Lip and/or Palate: Interventions and Return to Birth Weight. Cleft Palate Craniofac J. 2017 Mar;54(2):127-136. doi: 10.1597/15-163. Epub 2016 Feb 16. PMID 26882024
- [Background] Lao LJ, Zhang LY, DU LZ. [Malnutrition in early life and cardiovascular disease in adulthood]. Zhejiang Da Xue Xue Bao Yi Xue Ban. 2015 May;44(3):349-53. doi: 10.3785/j.issn.1008-9292.2015.05.18. Chinese. PMID 26350019
- [Background] Marques IL, Nackashi JA, Borgo HC, Martinelli AP, Pegoraro-Krook MI, Williams WN, Dutka JC, Seagle MB, Souza TV, Garla LA, Neto JS, Silva ML, Graciano MI, Moorhead J, Piazentin-Penna SH, Feniman MR, Zimmermann MC, Bento-Goncalves CG, Pimentel MC, Boggs S, Jorge JC, Antonelli PJ, Shuster J. Longitudinal study of growth of children with unilateral cleft-lip palate from birth to two years of age. Cleft Palate Craniofac J. 2009 Nov;46(6):603-9. doi: 10.1597/08-105.1. Epub 2009 May 16. PMID 19860503
- [Background] Martin V, Greatrex-White S. An evaluation of factors influencing feeding in babies with a cleft palate with and without a cleft lip. J Child Health Care. 2014 Mar;18(1):72-83. doi: 10.1177/1367493512473853. Epub 2013 Feb 25. PMID 23439590
- [Background] Montagnoli LC, Barbieri MA, Bettiol H, Marques IL, de Souza L. Growth impairment of children with different types of lip and palate clefts in the first 2 years of life: a cross-sectional study. J Pediatr (Rio J). 2005 Nov-Dec;81(6):461-5. doi: 10.2223/JPED.1420. PMID 16385363
- [Background] Pandya AN, Boorman JG. Failure to thrive in babies with cleft lip and palate. Br J Plast Surg. 2001 Sep;54(6):471-5. doi: 10.1054/bjps.2001.3618. PMID 11513506
- [Background] Ranalli DN, Mazaheri M. Height-weight growth of cleft children, birth to six years. Cleft Palate J. 1975 Oct;12:400-4. PMID 1058750
- [Background] Sawaya AL, Martins PA, Grillo LP, Florencio TT. Long-term effects of early malnutrition on body weight regulation. Nutr Rev. 2004 Jul;62(7 Pt 2):S127-33. doi: 10.1111/j.1753-4887.2004.tb00082.x. PMID 15387478
- [Background] Seth AK, McWilliams BJ. Weight gain in children with cleft palate from birth to two years. Cleft Palate J. 1988 Apr;25(2):146-50. PMID 3163290
- [Background] Smedegaard L, Marxen D, Moes J, Glassou EN, Scientsan C. Hospitalization, breast-milk feeding, and growth in infants with cleft palate and cleft lip and palate born in Denmark. Cleft Palate Craniofac J. 2008 Nov;45(6):628-32. doi: 10.1597/07-007.1. PMID 18956929
- [Background] Strupp BJ, Levitsky DA. Enduring cognitive effects of early malnutrition: a theoretical reappraisal. J Nutr. 1995 Aug;125(8 Suppl):2221S-2232S. doi: 10.1093/jn/125.suppl_8.2221S. PMID 7542704
- [Background] Young A. Cleft lip and/or palate. Community Pract. 2009 Jul;82(7):34-5. No abstract available. PMID 19626753